CLINICAL TRIAL: NCT01374165
Title: A Phase I Open Label, Unblinded, Single Dose Study for Evaluating the Safety and Pharmacokinetics of SANGUINATE™ in Sickle Cell Disease (SCD) Patients
Brief Title: Safety and Pharmacokinetics of SANGUINATE™ in Sickle Cell Disease (SCD) Patients
Status: Withdrawn | Type: Observational
Why Stopped: Study cancelled.
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SCIL-SANG-001
Record Dates: First submitted 2011-05-26; First posted 2011-06-15 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2015-01

CONDITIONS: Sickle Cell Disease
Keywords: SCD
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low dose SANGUINATE™: 160 mg/kg of SANGUINATE™.
  SANGUINATE™ (PEG-bHb-CO) an OTA is composed of three moieties, polyethylene glycol, bHb and carbon monoxide that act in a specific manner to promote the delivery of oxygen to tissue. SANGUINATE™ was not developed to be used as a blood substitute. It is instead an oxygen transfer agent intended to functionally deliver and release oxygen to hypoxic tissues.
- High dose of SANGUINATE™: 320 mg/kg of SANGUINATE™.
  SANGUINATE™ (PEG-bHb-CO) an OTA is composed of three moieties, polyethylene glycol, bHb and carbon monoxide that act in a specific manner to promote the delivery of oxygen to tissue. SANGUINATE™ was not developed to be used as a blood substitute. It is instead an oxygen transfer agent intended to functionally deliver and release oxygen to hypoxic tissues.

SUMMARY:
Prolong proposes to test safety, tolerability and pharmacokinetics of SANGUINATE™ in sickle cell disease (SCD) patients. Prolong's preclinical studies showed that SANGUINATE™ was safe in a number of different animal models and toxicology studies. In this Phase I trial, Prolong will test whether it is also safe and tolerable in sickle cell patients. The study will be conducted in 15 adult (>18 years) patients.

DETAILED DESCRIPTION:
This Phase I trial will test two doses of SANGUINATE™ in adult subjects suffering from chronic sickle cell disease (SCD). A total of fifteen (15) patients will be assigned to the low and high dose cohorts of SANGUINATE™.

The first 8 subjects will receive the study agent in an initial low dose of 160 mg/kg of SANGUINATE™.

Upon completion of the low dose cohort, safety variables will be reviewed by the Principal Investigator, the Study Manager, and the Sponsor (or designee) in order to determine the progression towards administration of a high dose cohort of 320 mg/kg of SANGUINATE™. 7 subjects will be enrolled in the high dose cohort. Subjects will not be enrolled in the next higher dose cohort until the dose in the preceding dose group is deemed safe and tolerable.

Sample Size: A total of 15 patients will be enrolled in the study (8 patients in the low dose cohort, 7 patients in the high dose cohort). In both cohorts an additional participant would not be enrolled prior to safety review of the results of the previously enrolled participant.

Dose and Mode of Administration: SANGUINATE™ is PEGylated bovine hemoglobin (PEG-Hb) in the CO form formulated in saline (PEG-Hb-CO).

The study drug is supplied in a 500 mL bag which is a red color sterile solution ready for infusion without any dilution or mixing.

SANGUINATE™ will be infused intravenously over 2 hours. The concentration of product is 40 mg/ml.

Dosing Schedule: The study will include two cohorts of SANGUINATE™:

The low dose cohort will receive 160 mg/kg; The high dose cohort will receive 320 mg/kg.

Laboratory and clinical assessments of each participant will be conducted during 24 hours (+/-1 hour) after the start of study drug administration. An additional participant would not be enrolled prior to safety review of the results of the previously enrolled participant in each cohort.

Upon completion of the low dose cohort, safety data will be reviewed by the Principal Investigator, Study Manager, and the Sponsor (or designee) in order to determine the progression towards administration of a high dose cohort.

Assessments:

Safety:

The following assessments will be used to evaluate the safety of SANGUINATE™ administration:

* adverse events, serious adverse events
* laboratory abnormalities by highest toxicity grade

A complete CBC with platelets will be performed at screening and Day 1 (upon admission to the clinical unit prior to dosing), and post-dose on Days 2, 3 and 7. Blood biochemistry testing (including amylase and lipase), and urinalysis with microscopic, will be performed at screening and Day 0 (admission), on Day 1 (6 hours post-infusion) and on Days 2, 3, 4, 5, and 7. Troponin I testing (cardiac assessment) will be performed at the discretion of PI upon Day 0 (admission), on Day 1 (baseline, 1, 3, and 6 hours post-infusion) and on Days 2, 3, 4, 5, and 7. Renal injury will be assessed via urinalysis and the following serum chemistry components: urea nitrogen, creatinine, creatinine clearance, potassium, chloride, magnesium and calcium. Pulse oximetry and arterial blood pressure will be captured on Day 1 at baseline, every 5 minutes during infusion, every 15 minutes post-infusion for 1 hour, and every 15 minutes thereafter until values return to baseline. Continuous 3-lead ECG monitoring will be performed on Day 1 from 15-min prior to infusion through 1 hour post-infusion and afterward until parameters return to baseline. 12-lead ECG will be captured at screening, Day 1 (baseline, immediately post-infusion, 10 hours post-infusion), and Days 2, 3 and 7.

Pharmacokinetics:

Descriptive statistics (N, mean, standard deviation, standard error of the mean, CV, median, minimum, and maximum) will be used to summarize single dose serum SANGUINATE™ concentration data at each planned sampling time point for both treatment cohort. Serial blood samples for pharmacokinetic analysis will be collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours from the start of infusion. Plasma will be analyzed by Prolong for concentrations of SANGUINATE™.

The blood volume required to perform the blood test for pharmacokinetic analysis is 5 ml at each collection time point.

Safety analyses will be performed and all adverse events and abnormal laboratory values will be assessed according to a standard grading system that will be provided. All safety analyses will be performed on the intent to treat population (all patients having received at least one dose and having at least one post baseline safety measurement). All data will be reported in individual patient listings.

Non-compartmental pharmacokinetic methods will be used to determine the pharmacokinetic parameter estimates of SANGUINATE™, which will include Cmax, Cmin, tmax, AUC 0->t, AUC 0 -> , t 1/2, CL/F, and accumulation index at steady state.

Precautionary Statement: Subjects must be informed that they may receive either low or high dose of drug SANGUINATE™ and that SANGUINATE™ has not been proven to be efficacious and safe in humans.

Possible Risks and Side Effects:

There are potential side effects resulting from the physical intravenous administration of any drug such as stinging, discomfort, bleeding, bruising, erythema or edema of the skin at the site of penetration and infusion.

Bovine hemoglobin has the potential to induce allergic responses, although SANGUINATE™ is designed specifically to reduce the likelihood of such symptoms. Symptoms that may be encountered in SANGUINATE™-allergic subjects include:

* Local skin reactions such as a wheal and flare response and local vascular reactions such as phlebitis.
* Wheezy breathlessness 1-7 hours after administration
* An increase in asthmatic symptoms.
* Rarely, anaphylactic responses may be encountered.

The bovine hemoglobin used for the manufacture of SANGUINATE™ has been purified to inactivate viruses and remove foreign proteins. There is no known risk for BSE/TSE.

ELIGIBILITY:
Eligibility Criteria:

Sickle cell patients will be enrolled and will be selected based on:

Inclusion:

1. Patients must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.
2. Hb levels: > 6 gr/dl - <10 gr/dl;
3. Age: > 18 - 65 years;
4. Body Mass Index ≥20 and ≤30 kg/m2;
5. Documented 12-lead ECG with no clinically significant abnormalities, as determined by the Investigator;
6. Female subjects of reproductive potential must have a negative serum pregnancy (β-HCG) test at screening and a negative urine pregnancy test at Day 0 prior to dosing. Female subjects must also be non-lactating;
7. Adequate venous access and can receive intravenous infusions;
8. Frequency of ER hospitalizations < 6x/yr for SCD pain events documented "medical history".

Exclusion:

1. In medical opinion of investigator, the patient is not an appropriate candidate;
2. Patient is infected;
3. The patient is Febrile;
4. Patient has Acute chest syndrome or documented Sickle Cell Crisis;
5. Patient with hemoglobin above 10gr/dl or below 6 gm/dl
6. If female, pregnant or lactating;
7. History of clinically significant disease, as determined by the Investigator;
8. History of allergy or major allergic reaction considered to be clinically significant by the Investigator;
9. Physical examination or 12-lead ECG result(s) considered to be clinically significant by the Investigator;
10. Received or intending to receive a vaccination in the two weeks prior to dosing, or anytime during study participation;
11. Unable to comply with study attendance, protocol procedures or other study requirements;
12. Frequency of ER hospitalizations > 6x/yr for SCD pain events;
13. Patient has Renal or liver dysfunction;
14. Patient has Severe pulmonary hypertension (index > 3 meters per sec based on documented Echocardiograph);
15. Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results;
16. Screening laboratory result indicating HIV-positivity, or previously diagnosed with AIDS, AIDS related complex, or other immunodeficiency;
17. Screening laboratory result indicating serologic positivity for hepatitis C antibodies or hepatitis B surface antigens, unless explained by a documented vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sickle Cell Disease (SCD) patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of two dose regimen for SANGUINATE™ in sickle cell disease patients | 7 days
  The following assessments will be used to evaluate the safety of SANGUINATE™ administration:
  * adverse events, serious adverse events
  * laboratory abnormalities by highest toxicity grade
  * laboratory abnormalities by largest increase in toxicity grade from baseline

SECONDARY OUTCOMES:
Determine the plasma pharmacokinetic (PK) profile of SANGUINATE™ in sickle cell disease patients. Mean values by treatment received will be calculated for the following PK parameters for PEGylated bovine hemoglobin: | 7 Days
  * Cmax -the maximum measured plasma concentration
  * tmax -the time to reach maximum plasma concentration
  * AUC0-last -the area under the plasma concentration versus time curve from time zero to the time of the last measurable plasma concentration, calculated by the linear or log/linear trapezoidal method
  * AUC0-inf -the area under the plasma concentration versus time curve from time zero to infinity, calculated as: AUCinf = AUCt + (Ct/Kel), where Ct = the last measurable concentration
  * λz -the apparent elimination rate constant
  * t1/2 -the terminal half-life
  * CV -coefficient of variation

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Acharya AS, Intaglietta M., Tsai AG, Malavalli A., Vandegriff K., Winslow RM, Smith PK, Friedman JM, and Manjula BN. Enhanced molecular volume of conservatively PEGylated Hb: (SP-PEG5K).sub.6-HbA is non-hypertensive. Artificial cells, Blood Subs. Biotechnol. 2005; 33: 239-255 Atochin DN, Wang A., Liu VW, Critchlow JD, Dantas AP, Looft-Wilson R., Murata T., Salomone S., Shin HK, Ayata, C., Moskowitz MA, Michel T., Sessa WC, Huang PL. The phosphorylation state of eNOS modulates vascular reactivity and outcome of cerebral ischemia in vivo. J Clin Invest. 2007 Jul; 117(7):1961-7. Cao S., Wang L-C, Kwansa, H., Roman RJ, Harder DR, Koehler RC. Endothelin rather than 20-HETE contributes to loss of pial arteriolar dilation during focal cerebral ischemia without polymeric hemoglobin transfusion. Am J Physiol Regulatory Integr ative Comp Physiol. 2009 May; 296(5):R1412-8. Castro O, Management of Sickle Cell Disease: Recent advances and controversies. Brit J. of Hematology. 1999 Oct; 2-11 Conover CD, Linberg R., Shum KL, Shorr RG. The ability of polyethylene glycol conjugated bovine hemoglobin (PEG-Hb) to adequately deliver oxygen in both exchange transfusion and top-loaded rat models. Artif. Cells Blood Substit. Immobil. Biotechnol. 1999; 27:93-107 Gould SA, Moore EE, Hoyt DB, Burch JM, Haenel JB, Garcia J., DeWoskin R, Moss GS: The first randomized trial of human polymerized hemoglobin as a blood substitute in acute trauma and emergent surgery. J Am Coll Surg. 1998;187:113-120. Gould SA, Moore EE, Hoyt DB, Ness PM, Norris EJ, Carson JL, Hides GA, Freeman IH, DeWoskin R., Moss GS: The life-sustaining capacity of human polymerized hemoglobin when red cells might be unavailable. J Am Coll Surg 2002; 195:445-52; discussion 452-5 Koehler RC, Traystman RJ. Cerebrovascular effects of carbon monoxide. Antioxidants and Redox Signaling 4: 279-290, 2002